CLINICAL TRIAL: NCT05803707
Title: Home-based Adapted Physical Activity in Anorexia Nervosa: a Feasibility Pilot Study
Acronym: APAMAdom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC22.0097
Record Dates: First submitted 2022-12-23; First posted 2023-04-07 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; telerehabilitation; Adapted Physical Activity
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Adapted Physical Activity (Experimental): Home-based Adapted Physical Activity sessions by videoconference
  Interventions: Behavioral: Home-based Adapted Physical Activity

INTERVENTIONS:
Behavioral: Home-based Adapted Physical Activity — There will be 8 weekly sessions at a time defined in advance for the same group and for the 8 sessions

SUMMARY:
The goal of this pilot clinical trial is to assess a program of Home-based Adapted Physical Activity in Anorexia Nervosa.

DETAILED DESCRIPTION:
The main questions it aims to answer are: Determining the acceptability of this program / Determining the feasibility and safety of this program / Determining patient satisfaction / Measuring the evolution of the symptomatology. Participants will follow a program of Home-based Adapted Physical Activity.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 18 and 60 years
* Subjects able to give informed consent
* Eating disorders such as anorexia nervosa
* BMI < 18.5 kg/m2
* Affiliated in a social security plan
* Having given informed consent to the research

Exclusion Criteria:

* Indication for in-patient care or BMI < 12 kg/m2
* Subject presenting a contrindication to the practice of an adapted physical activity
* Anorexia nervosa in partial or complete remission for more than 1 year
* Patient unable, for technical or any other reason, to connect via the Internet for tele-monitoring and/or tele-rehabilitation
* Persons concerned by the articles L1121-5 to L1121-8 of the public health code
* Subjects who cannot be contacted in case of emergency
* Subjects in a period of exclusion from another study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of a telerehabilitation adapted physical activity (APA) program for patient with anorexia nervosa quantitatively | at the first session of the APA program (Day 0)
  Number of patients who have realized the first of the 8 adapted physical activity session in relation to the total number of eligibly patients who have been invited to participate at the study
Acceptability of a telerehabilitation adapted physical activity program for patient with anorexia nervosa qualitively | at the first session of the APA program (Day 0)
  Reasons for refusal and participation's age will be collected anonymously for patients who refuse inclusion but agree to this informations being collected
Feasibility and safety of a telerehabilitation adapted physical activity program for patients with anorexia nervosa quantitatively | at the end-of-study visit (Day 0 + 11 weeks)
  Number and portion of patients who have realized the 8 adapted physical activity sessions as well as the first and final sessions
Feasibility and safety of a telerehabilitation adapted physical activity program for patients with anorexia nervosa qualitively | at the end-of-study visit (Day 0 + 11 weeks)
  Motifs of no realization of one ou more sessions will be collected. They will inclued technical problems, personal, professional ou medical constraints inclued study's exit for weight loss
Patient satisfaction with the telerehabilitation adapted physical activity program for patients with anorexia nervosa quantitatively | at the final session of APA programm (Day 0 + 8 weeks)
  Portion of patients answing "yes" at the question : "Would you like to continue this program ?"
Patient satisfaction with the telerehabilitation adapted physical activity program for patients with anorexia nervosa qualitively | at the final session of APA programm (Day 0 + 8 weeks)
  Programm's motifs of satisfaction or no satisfaction will be collected during the final session of adapted physical activity program
Measuring changes in symptomatology in key areas such as self-esteem through self-assessment questionnaire | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parameter :self-esteem by self-esteem scale of Rosenberg
Measuring changes in symptomatology in key areas such as quality of life through self-assessment questionnaire | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parametes :quality of life by QUAVIAM scale
Measuring changes in symptomatology in key areas such as dependence on physical activity through self-assessment questionnaire | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parameter : dependence on physical activity by EDQ questionnary
Measuring changes in symptomatology in key areas such as dependence on physical activity through objective measure | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parameter : level of physical activity by 7-day actimetry recording
Measuring changes in symptomatology in key areas such as changes in weight through objective measure | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parameter : weight in kilograms on a classic scale
Measuring changes in symptomatology in key areas such as body composition through objective measure | at the early study visit (Day 0 - 4 weeks) and at end-of-study visit (Day 0 + 11 weeks )
  Determination of this parameters : the body composition will be determinated by a impedancemetry measurement

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cécile BETRY, Grenoble
  - Pr GUILLAUME Sébastien, Montpellier